CLINICAL TRIAL: NCT05785520
Title: Evaluation of the Effect on Functionality of the "ST500 SINGLE- DOSE GEL" Medical Device in Patients With Symptomatic Long Head of the Biceps Tendon Injury: a Postmarket Interventional, Single Arm Clinical Investigation
Brief Title: Evaluation of the "ST500 SINGLE- DOSE GEL" in Patients With Symptomatic Long Head of the Biceps Tendon Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Contrad Swiss SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTD-SW ST500
Record Dates: First submitted 2023-02-21; First posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-02

CONDITIONS: Long Head of Biceps Rupture
Keywords: Long Head of Biceps; Long Head of Biceps Tendon Injury; Hyaluronic Acid; Peptides; LHBT injury; Constant-Murley Score

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ST500 single-dose gel (Other): The treatment is performed twice weekly for 6 weeks.
  Interventions: Device: ST500 SINGLE-DOSE GEL

INTERVENTIONS:
Device: ST500 SINGLE-DOSE GEL — ST500 SINGLE-DOSE GEL is a hydrogel to be applied to intact skin, useful to limit the physiological degeneration of the joints and tissues, improving their functionality. The presence of a peptide mixture and sodium hyaluronate facilitates the movement of joints and tendons for greater mobility and flexibility.

SUMMARY:
Single arm, post-market, confirmatory, interventional clinical investigation - Medical Device

DETAILED DESCRIPTION:
The aim of this single arm, post-market, confirmatory, interventional clinical investigation was to evaluate the effect on shoulder functionality and symptoms in patients affected by LHBT injury of a HA-based gel containing a peptide mixture, the ST500 SINGLE-DOSE GEL (ST500TM), topically applied to the shoulder.

ELIGIBILITY:
Inclusion Criteria:

1. Male or Female, aged ≥18 years at the time of the signature of ICF.
2. Unilateral or bilateral LHBT injury of mild or moderate severity (CMS ≤ 70).
3. Willing to follow all study procedures, including attending all site visits, tests and examinations.
4. Willing to participate in the study and sign the ICF.

Exclusion Criteria:

1. Other - different - clinical conditions of the shoulder requiring surgical intervention as well as full rotator cuff tears and LHBT lesions classified as Type IV, V, or VI.
2. Previous shoulder(s) surgery.
3. Infective or inflammatory processes near the area of treatment.
4. Damaged skin in the area of treatment.
5. Ongoing cutaneous allergies.
6. Serious and chronical pathological skin conditions (i.e., rosacea, psoriasis, vitiligo) including diagnosticated cancer with/without ongoing antitumor therapy.
7. Allergy to device components (Sodium hyaluronate; SH-Polypeptide-29; SH-Tripeptide-1; Demineralized water; Glycerin; Propylene glycol; Ethylhexylglycerin; Panthenol; PEG-40 hydrogenated castor oil; Sodium hydroxide; Xanthan gum; Phenoxyethanol; Benzoic Acid; Carbomer; Dehydroacetic Acid; Disodium EDTA).
8. Any other systemic or local therapy for the treatment of LHBT injury (only physiotherapy is allowed).
9. Any other systemic or local therapy (e.g. corticosteroids) for the treatment of other inflammatory diseases (e.g. dermatitis, acute or chronic bronchitis, gastroenteritis, etc.) or painful states (e.g. headache, dental abscess, etc.) that may interfere with the clinical course of LHBT injury under treatment with the medical device ST500 (only the use of paracetamol, according the procedures described in the protocol, is allowed to treat the painful state related to LHBT injury).
10. High consumption of analgesic drugs for the painful state upon clinician judgement (i.e., NSAIDs + opioid or NSAIDs + steroids).
11. Immune system illnesses.
12. Uncontrolled systemic diseases.
13. Known drug and/or alcohol abuse.
14. Mental incapacity that precludes adequate understanding or cooperation.
15. Participation in another investigational study.
16. Pregnancy or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2021-11-30 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2022-10-10 (Actual)

PRIMARY OUTCOMES:
Clinical performance of the ST500™ in the increase of shoulder functionality, in terms of difference (percent) in the Constant-Murley Score (CMS) between the end of study visit and baseline visit. | 10 weeks
  To evaluate the clinical performance of the ST500™ in the increase of shoulder functionality, in terms of difference (percent) in the Constant-Murley Score (CMS) between the end of study visit and baseline visit, in patients affected by Long Head of the Biceps Tendon (LHBT) injury.
  The Constant-Murley score (CMS) is a 100-points scale, that ranges from 0 points (most disability) to 100 points (least disability).

SECONDARY OUTCOMES:
Clinical performance of the ST500™ in supporting the physiological regenerative process of tendon | 10 weeks
  To evaluate the clinical performance of the ST500™ in supporting the physiological regenerative process of tendon assessed by high resolution ultrasound (HRUS)
Clinical performance of the ST500 in the attenuation of disability in patients affected by LHBT injury | 10 weeks
  To evaluate the clinical performance of the ST500 in the attenuation of disability in patients affected by Long Head of the Biceps Tendon (LHBT) injury assessed by range of motion through use of a digital goniometer.
Number of participants with Adverse Events (ST500 Safety and Tolerability) | 10 weeks
  To evaluate the tolerability and safety of ST500™ through identification of Adverse Events including assessment of the relationship of the Adverse Event to the Investigational Product (e.g. local allergic reaction).
Patient satisfaction of the ST500™ | 10 weeks
  To evaluate the tolerability and patient satisfaction of the CR 500™ through a the completion of a specific questionnaire by the patient, the five-points Likert scale in which 1 means Strongly disagree with the assertion and 5 means Strongly agree

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Luini Confalonieri, Luino, Varese, Italy

IPD SHARING:
Plan to Share IPD: Undecided